CLINICAL TRIAL: NCT05317897
Title: Utility of Lung Ultrasonography As a Predictor of Fast Track Extubation in Pediatric Cardiac Surgeries an Observational Study
Brief Title: Utility of Lung Ultrasonography As a Predictor of Fast Track Extubation
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Lecturer of Anesthesia, ICU and Pain managment, Kasr El Aini Hospital
Other Study IDs: MS-235-2017
Record Dates: First submitted 2022-03-25; First posted 2022-04-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Exta Vascular Lung Water

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound examination — 45 pediatric patients who will go elective repair of congenital acyanotic heart diseases will be included and will be examined with Lung ultrasound together with arterial blood gases preoperative and postoperative and given a score range from 0-3 according to number of B lines in each region and sensitivity of post-operative lung ultrasound score to extubation within 6 hours was examined.
  Other Names: The lung ultrasound score

SUMMARY:
Fast-tracking in cardiac surgery refers to early extubation to reduce costs and perioperative morbidity. The use of lung ultrasound is recently accepted as a tool in the assessment of several lung conditions. The aim of this study was to assess the use of lung ultrasound score as a quantitative method to assist in the decision of early extubation.

DETAILED DESCRIPTION:
background: Fast-tracking in cardiac surgery refers to early extubation to reduce costs and perioperative morbidity. The use of lung ultrasound is recently accepted as a tool in the assessment of several lung conditions. The aim of this study was to assess the use of lung ultrasound score as a quantitative method to assist in the decision of early extubation.

Methedology: in this prospective, observational study, 45 pediatric patients who will go elective repair of congenital acyanotic heart diseases were included and were examined with Lung ultrasound together with arterial blood gases preoperative and postoperative and given a score range from 0-3 according to number of B lines in each region and sensitivity of post-operative lung ultrasound score to extubation within 6 hours was examined Demographic data: Patients' name, age, sex, diagnosis, relevant medical and surgical history. And Assessment data: Baseline arterial blood gases and lung ultrasound score assessment after induction of anesthesia and at the end of surgery.

Primary outcome will be the sensitivity of lung ultrasound scores immediately at the end of pediatric cardiac operation in prediction of extubation. and Secondary outcome will be correlation between lung ultrasound score and Po2/Fio2 ratio at the end of operation

ELIGIBILITY:
Inclusion Criteria:

* were Age 6 months to 7 years
* Patients suffering from Acyanotic congenital heart diseases.

Exclusion Criteria:

* Age is less than 6 months and more than 7 years,
* Preoperative mechanical ventilation,
* Preoperative inotropic support.,
* Trisomy 21,
* Patient with cyanotic heart diseases
* Coagulopathy INR >1.5

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients suffering from Acyanotic congenital heart diseases.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
the sensitivity of lung ultrasound scores | immediately at the end of pediatric cardiac operation
  the sensitivity of lung ultrasound scores immediately at the end of pediatric cardiac operation in prediction of extubation

SECONDARY OUTCOMES:
correlation between lung ultrasound score and Po2/Fio2 ratio | immediatly at the end of pediatric cardiac operation until 6 hours post operative until extubatiioon
  correlation between lung ultrasound score and Po2/Fio2 ratio at the end of operation

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kasr Al Ainy Hospital, Cairo, Cairo Governorate
  - Kasr Alainy hospital, Cairo

IPD SHARING:
Plan to Share IPD: No